CLINICAL TRIAL: NCT06261814
Title: 2D and 3D Contrast Enhanced Ultrasound of Chemoembolization
Brief Title: Contrast Enhanced Ultrasound to Evaluate Response to Chemoembolization in Patients With Liver Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: john eisenbrey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, john eisenbrey, Principal Investigator, Thomas Jefferson University
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: iRISID-2023-2142; JT 33825 (Other: JeffTrial Number); R01CA194307 (NIH)
Record Dates: First submitted 2024-02-07; First posted 2024-02-15 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-02

CONDITIONS: Liver Neoplasms
MeSH Terms: conditions — Liver Neoplasms | interventions — Chemoembolization, Therapeutic

STUDY DESIGN:
Intervention Model Description: No Data Available
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diagnostic (CEUS) (Experimental): Patients receive lumason IV and undergo CEUS 2 weeks prior to TACE, during TACE, 1-2 weeks after TACE, and then 1-2 months after TACE.
  Intervention(s)
  Interventions: Drug: Sulfur Hexafluoride Lipid Microspheres; Procedure: Contrast-Enhanced Ultrasound; Procedure: Transarterial Chemoembolization; Other: Medical Chart Review

INTERVENTIONS:
Drug: Sulfur Hexafluoride Lipid Microspheres — Given IV
  Other Names: Lumason; SF6 Lipid Microspheres; Sulfur Hexafluoride Lipid-type A Microspheres
Procedure: Contrast-Enhanced Ultrasound — Undergo CEUS
  Other Names: CEUS
Procedure: Transarterial Chemoembolization — Undergo TACE
  Other Names: TACE; Chemoembolization
Other: Medical Chart Review — Ancillary studies
  Other Names: Chart Review

SUMMARY:
This phase II trial evaluates the diagnostic performance of contrast-enhanced ultrasound (CEUS) for assessing treatment response in patients undergoing transarterial chemoembolization (TACE) for liver tumors. TACE is a hepatic artery embolization technique involving the injection of a blocking agent and a chemotherapy agent to treat liver cancers. Currently, contrast enhanced magnetic resonance imaging or computed tomography are used to assess disease response 1-2 months after TACE treatment, but ultrasound may be a less expensive, earlier alternative. CEUS is an imaging procedure that uses high-frequency sound waves to generate images of the body after administering Lumason, an imaging agent used to enhance visualization of blood flow on ultrasounds. CEUS is able to be performed during the TACE procedure, making it possible to evaluate treatment response earlier than standard techniques. CEUS may be an effective method to evaluate treatment response more accurately and much earlier than current standard evaluation methods.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the sensitivity and specificity of CEUS for the evaluation of TACE treatment response in a variety of solid liver tumors (years 1-4).

SECONDARY OBJECTIVES:

I. To determine the ability of CEUS to identify residual tumor vascularity intraoperatively, thereby enabling immediate retreatment when necessary (years 1-4).

II. To explore a variety of advanced imaging approaches to improve on the suboptimal specificity of CEUS for identifying residual viable tumor following TACE (years 1-5).

III. To investigate the ability of CEUS obtained prior to TACE to quantitatively assess tumor vascular morphology and predict response to therapy (years 2-5).

EXPLORATORY OBJECTIVE:

I. Use acquired B-mode in-phase and quadrature (IQ) data for H-scan imaging.

OUTLINE:

Patients receive sulfur hexafluoride lipid microspheres (Lumason) intravenously (IV) and undergo CEUS 2 weeks prior to TACE, during TACE, 1-2 weeks after TACE, and then 1-2 months after TACE.

After completion of study treatment, patients are followed up at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for TACE therapy of a liver tumor
* Be at least 18 years of age
* Be medically stable
* If a female of child-bearing age, must have a negative pregnancy test
* Have signed informed consent to participate in the study

Exclusion Criteria:

* Patients who are medically unstable, patients who are seriously or terminally ill, and patients whose clinical course is unpredictable
* Patients with known sensitivities to the components of lumason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Estimated)
Dates: Start 2024-08-07 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence | Up to 6 months
Sensitivity | Up to 6 months
  Will be computed using a reference standard. Variables will be summarized with descriptive statistics, such as means with standard deviations or frequency counts with percentage, across the cohort and within group of interest. Diagnostic accuracy will be compared between hepatocellular carcinoma (HCC) and non-HCC and between all tumor subtypes.
Specificity | Up to 6 months
  Will be computed using a reference standard. Variables will be summarized with descriptive statistics, such as means with standard deviations or frequency counts with percentage, across the cohort and within group of interest. Diagnostic accuracy will be compared between HCC and non-HCC and between all tumor subtypes.
Positive predictive value | Up to 6 months
  Will be computed using a reference standard. Variables will be summarized with descriptive statistics, such as means with standard deviations or frequency counts with percentage, across the cohort and within group of interest. Diagnostic accuracy will be compared between HCC and non-HCC and between all tumor subtypes.
Negative predictive value | Up to 6 months
  Will be computed using a reference standard. Variables will be summarized with descriptive statistics, such as means with standard deviations or frequency counts with percentage, across the cohort and within group of interest. Diagnostic accuracy will be compared between HCC and non-HCC and between all tumor subtypes.
False discovery rate | Up to 6 months
  Will be computed using a reference standard. Variables will be summarized with descriptive statistics, such as means with standard deviations or frequency counts with percentage, across the cohort and within group of interest. Diagnostic accuracy will be compared between HCC and non-HCC and between all tumor subtypes.

SECONDARY OUTCOMES:
Residual tumor vacularity | Up to 6 months
  Will use diagnostic summary statistics and generalized estimating equations (GEE) logistic regression modeling. The bedside (interventional radiologist) versus offline (radiologist) reads will be compared using agreement, kappa statistics, and mixed modeling.
Diagnostic performance for each imaging mode | Up to 6 months
  The diagnostic performance for each reader will be quantified from the volumetric contrast enhanced ultrasound exams and post-processed images. Diagnostic performance for each imaging mode will be compared across all readers using the GEE logistic regression approach. Quantitative H-scan data will be compared between complete and incomplete responders using multiple linear regression or GEE regression modeling, depending on how well assumptions hold for the former.
Ability of the model to predict binary treatment response | Up to 6 months
  Model performance will be calculated using a leave-one-out cross-validation method to assess the ability of the model to predict binary treatment response. Accuracy, sensitivity and specificity will then be quantified and directly compared between 2 dimensional (D) and 3D datasets.

CONTACTS AND LOCATIONS:
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States